CLINICAL TRIAL: NCT00008372
Title: Phase II Trial Of CQS (NSC 339004) In Platinum-Refractory Small Cell Lung Cancer
Brief Title: Chloroquinoxaline Sulfonamide in Treating Patients With Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: 00104; P30CA033572 (NIH); CHNMC-PHII-26; NCI-57; CDR0000068401 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 2001-01-06; First posted 2003-11-11 (Estimated); Last update posted 2011-10-20 (Estimated); Status verified 2011-10

CONDITIONS: Lung Cancer
Keywords: extensive stage small cell lung cancer; recurrent small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Small Cell Lung Carcinoma | interventions — 5-chloroquinoxaline-2-sulfanilamide

INTERVENTIONS:
Drug: chloroquinoxaline sulfonamide

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of chloroquinoxaline sulfonamide in treating patients who have small cell lung cancer that has not responded to platinum-based chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the efficacy of chloroquinoxaline sulfonamide in patients with platinum-refractory small cell lung cancer. II. Determine the toxic effects of this drug in these patients.

OUTLINE: Patients receive chloroquinoxaline sulfonamide IV over 1 hour once a week for 4 weeks. Treatment repeats every 6 weeks in the absence of disease progression or unacceptable toxicity. Patients are followed until death.

PROJECTED ACCRUAL: A total of 12-38 patients will be accrued for this study within 12-18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed platinum-refractory small cell lung cancer No response or progression during or within 6 months of completing platinum based therapy Measurable disease No symptomatic brain or leptomeningeal metastases

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: SWOG 0-2 Life expectancy: At least 12 weeks Hematopoietic: Granulocyte count at least 1,500/mm3 Platelet count at least 100,000/mm3 No hemolytic anemia Hepatic: Bilirubin normal AST no greater than 2.5 times upper limit of normal Renal: Creatinine no greater than 1.5 mg/dL OR Creatinine clearance at least 60 mL/min Cardiovascular: No history of cardiac arrhythmias Other: No other active malignancy requiring concurrent treatment No allergy to sulfonamides Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: See Disease Characteristics No more than 2 prior chemotherapy regimens At least 3 weeks since prior chemotherapy and recovered Endocrine therapy: No concurrent corticosteroids to control symptoms of brain and/or leptomeningeal metastases Radiotherapy: At least 4 weeks since prior radiotherapy No concurrent radiotherapy to measurable lesions Surgery: Not specified Other: No concurrent hypoglycemic agents (including insulin)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-12; Primary Completion 2002-09 (Actual); Study Completion 2002-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Primo N. Lara, MD, Study Chair — University of California, Davis
Locations (3):
- United States (3):
  - Cancer Center and Beckman Research Institute, City of Hope, Duarte, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - University of California Davis Cancer Center, Sacramento, California